CLINICAL TRIAL: NCT05352698
Title: Validation of B-type Natriuretic Peptide With N-terminal Pro B-type Natriuretic Peptide in Perioperative Risk Assessment
Status: Completed | Type: Observational
Sponsor: Jordan Leitch (Other)
Responsible Party: Sponsor-Investigator, Jordan Leitch, Principal Investigator, Queen's University
Organization: Queen's University (Other)
Other Study IDs: 6035639
Record Dates: First submitted 2022-04-19; First posted 2022-04-29 (Actual); Last update posted 2024-06-24 (Actual); Status verified 2024-06

CONDITIONS: Perioperative Care
Keywords: BNP; NT ProBNP; MINS; myocardial injury after non-cardiac surgery; perioperative risk; risk stratification; perioperative care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Non-Cardiac Surgery Patient: Our study population will be comprised of any patient undergoing non-cardiac surgery who meets standard of care criteria for BNP testing. This includes patients who are a) >65 years old, b) revised cardiac risk index (RCRI) ≥1 or c) >45 years old with significant cardiovascular disease (coronary artery disease, peripheral arterial disease, cerebral vascular disease, congestive heart failure, obstructive intracardiac disease such as severe aortic stenosis, severe mitral stenosis or severe hypertrophic obstructive cardiomyopathy)
  Interventions: Diagnostic Test: NT ProBNP (Roche)

INTERVENTIONS:
Diagnostic Test: NT ProBNP (Roche) — This NT ProBNP assay is a point-of-care (POC) test that will be conducted on a 2 mL sample of whole blood collected in a non-heparinized tube. NT ProBNP results are used in this setting to predict perioperative cardiovascular risk.

SUMMARY:
This is a single-centre, prospective study to determine the correlation and comparative thresholds between N-terminal pro-brain natriuretic peptide (NT ProBNP, Roche) and brain natriuretic peptide (BNP, Abbott) tests. The study population will include patients assessed in presurgical screening (PSS) or on the day of surgery (DOS) who are presenting for elective surgery requiring a minimum of one-night admission, and are a) >65 years old, b) RCRI ≥1 or c) >45 years old with significant cardiovascular disease (coronary artery disease, peripheral arterial disease, cerebral vascular disease, congestive heart failure, obstructive intracardiac disease such as severe aortic stenosis, severe mitral stenosis or severe hypertrophic obstructive cardiomyopathy). Informed consent will be obtained at PSS or on the DOS by study staff. High sensitivity troponin I measurements will be taken on postoperative day (POD) 0, 1 and 2, and the outcome of MINS (high sensitivity troponin > 30 ng/L) or vascular death will be determined by an assessor blinded to BNP/NT ProBNP results at postoperative day (POD) 30. Given a sample size of 431 patients and based upon previous local data that found approximately 500 patients qualifying for BNP testing in a six month period, the investigators predict data collection to be completed in approximately six months.

DETAILED DESCRIPTION:
This is a single-centre, prospective study to determine the correlation and comparative thresholds between NT ProBNP (Roche) and BNP (Abbott) tests. This will involve simultaneous serum sampling for both BNP and NT ProBNP at pre-surgical screening (PSS) or on the day of surgery (DOS). Serum sampling of BNP in this patient population is standard of care in our institution, thus only the additional blood required for the NT ProBNP test requires additional consent. Informed consent will be obtained at PSS or on the DOS by study staff. High sensitivity troponin I (Abbott) measurements will be taken on postoperative day (POD) 0, 1 and 2, as per local standard of care and the outcome of MINS (myocardial injury after non-cardiac surgery as indicated by high sensitivity troponin > 30 ng/L) or vascular death will be determined by an assessor blinded to BNP/NT ProBNP results at postoperative day (POD) 30. The primary outcome is correlation of POC NT ProBNP with BNP levels and validation of appropriate thresholds. The secondary outcome is combined MINS and vascular death at POD 30.

The study population will include patients assessed in PSS or on the DOS who are presenting for elective surgery requiring a minimum of one-night admission following and are a) >65 years old, b) revised cardiac risk index (RCRI) ≥1 or c) >45 years old with significant cardiovascular disease (coronary artery disease, peripheral arterial disease, cerebral vascular disease, congestive heart failure, obstructive intracardiac disease such as severe aortic stenosis, severe mitral stenosis or severe hypertrophic obstructive cardiomyopathy).

The required sample size of 431 patients was calculated to adequately perform a power assessment of the primary outcome of correlating BNP and NT ProBNP thresholds. Historically, Presurgical Screening (PSS) at Kingston Health Sciences Centre (KHSC) collects BNP serum samples from approximately 500 patients at PSS in a six month time frame, as reported by a local, retrospective quality assurance study (McMullen/Cook). This sample size will not likely be sufficient to determine significance regarding the secondary outcome of MINS or vascular death by POD 30. Nonetheless, the trend observed may be informative in the context of correlating the risk prediction provided by BNP screening at our centre to that from larger studies.

ELIGIBILITY:
Inclusion Criteria:

* Patient consents to study and is undergoing non-cardiac surgery and is one of:
* Age > 65 years
* Revised cardiac risk index (RCRI) >=1
* Age > 45 years old with significant cardiovascular disease (coronary artery disease, peripheral arterial disease, cerebral vascular disease, congestive heart failure, obstructive intracardiac disease such as severe aortic stenosis, severe mitral stenosis or severe hypertrophic obstructive cardiomyopathy)

Exclusion Criteria:

* Age < 18 years
* Patient undergoing cardiac surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will include patients assessed in pre-surgical screening or on the day of surgery who are presenting for non-cardiac surgery requiring a minimum of one-night admission following and are a) >65 years old, b) RCRI ≥1 or c) >45 years old with significant cardiovascular disease (coronary artery disease, peripheral arterial disease, cerebral vascular disease, congestive heart failure, obstructive intracardiac disease such as severe aortic stenosis, severe mitral stenosis or severe hypertrophic obstructive cardiomyopathy).
Sampling Method: Non-Probability Sample
Enrollment: 466 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
BNP/NT ProBNP Conversion Formula | Within three months before surgery
  The primary objective of this study is to determine external validation of the BNP (Abbott)/NT ProBNP conversion formula (Kasahara et al., 2019) and to provide recalibration, if necessary, for the POC NT ProBNP results.

SECONDARY OUTCOMES:
POD30 Myocardial injury after non-cardiac surgery (MINS) | 30 days after surgery
  Incidence of thirty-day post-operative myocardial injury after non-cardiac surgery (MINS) as determined by high-sensitivity troponin I (Abbott) > 30 ng/L
POD30 Vascular Death | 30 days after surgery
  Thirty day vascular death is defined as death from the composite of these vascular diseases: hypertensive disease, ischemic heart disease, cerebrovascular disease, pulmonary vascular disease, renal failure, artery/arteriole/capillary disease.

CONTACTS AND LOCATIONS:
Locations (1):
- Kingston Health Sciences Centre, Kingston, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP

REFERENCES:
- [Background] Writing Committee for the VISION Study Investigators; Devereaux PJ, Biccard BM, Sigamani A, Xavier D, Chan MTV, Srinathan SK, Walsh M, Abraham V, Pearse R, Wang CY, Sessler DI, Kurz A, Szczeklik W, Berwanger O, Villar JC, Malaga G, Garg AX, Chow CK, Ackland G, Patel A, Borges FK, Belley-Cote EP, Duceppe E, Spence J, Tandon V, Williams C, Sapsford RJ, Polanczyk CA, Tiboni M, Alonso-Coello P, Faruqui A, Heels-Ansdell D, Lamy A, Whitlock R, LeManach Y, Roshanov PS, McGillion M, Kavsak P, McQueen MJ, Thabane L, Rodseth RN, Buse GAL, Bhandari M, Garutti I, Jacka MJ, Schunemann HJ, Cortes OL, Coriat P, Dvirnik N, Botto F, Pettit S, Jaffe AS, Guyatt GH. Association of Postoperative High-Sensitivity Troponin Levels With Myocardial Injury and 30-Day Mortality Among Patients Undergoing Noncardiac Surgery. JAMA. 2017 Apr 25;317(16):1642-1651. doi: 10.1001/jama.2017.4360. PMID 28444280
- [Background] Vascular Events In Noncardiac Surgery Patients Cohort Evaluation (VISION) Study Investigators; Devereaux PJ, Chan MT, Alonso-Coello P, Walsh M, Berwanger O, Villar JC, Wang CY, Garutti RI, Jacka MJ, Sigamani A, Srinathan S, Biccard BM, Chow CK, Abraham V, Tiboni M, Pettit S, Szczeklik W, Lurati Buse G, Botto F, Guyatt G, Heels-Ansdell D, Sessler DI, Thorlund K, Garg AX, Mrkobrada M, Thomas S, Rodseth RN, Pearse RM, Thabane L, McQueen MJ, VanHelder T, Bhandari M, Bosch J, Kurz A, Polanczyk C, Malaga G, Nagele P, Le Manach Y, Leuwer M, Yusuf S. Association between postoperative troponin levels and 30-day mortality among patients undergoing noncardiac surgery. JAMA. 2012 Jun 6;307(21):2295-304. doi: 10.1001/jama.2012.5502. PMID 22706835
- [Background] Duceppe E, Parlow J, MacDonald P, Lyons K, McMullen M, Srinathan S, Graham M, Tandon V, Styles K, Bessissow A, Sessler DI, Bryson G, Devereaux PJ. Canadian Cardiovascular Society Guidelines on Perioperative Cardiac Risk Assessment and Management for Patients Who Undergo Noncardiac Surgery. Can J Cardiol. 2017 Jan;33(1):17-32. doi: 10.1016/j.cjca.2016.09.008. Epub 2016 Oct 4. PMID 27865641
- [Background] Duceppe E, Patel A, Chan MTV, Berwanger O, Ackland G, Kavsak PA, Rodseth R, Biccard B, Chow CK, Borges FK, Guyatt G, Pearse R, Sessler DI, Heels-Ansdell D, Kurz A, Wang CY, Szczeklik W, Srinathan S, Garg AX, Pettit S, Sloan EN, Januzzi JL Jr, McQueen M, Buse GL, Mills NL, Zhang L, Sapsford R, Pare G, Walsh M, Whitlock R, Lamy A, Hill S, Thabane L, Yusuf S, Devereaux PJ. Preoperative N-Terminal Pro-B-Type Natriuretic Peptide and Cardiovascular Events After Noncardiac Surgery: A Cohort Study. Ann Intern Med. 2020 Jan 21;172(2):96-104. doi: 10.7326/M19-2501. Epub 2019 Dec 24. PMID 31869834
- [Background] Farnsworth CW, Bailey AL, Jaffe AS, Scott MG. Diagnostic concordance between NT-proBNP and BNP for suspected heart failure. Clin Biochem. 2018 Sep;59:50-55. doi: 10.1016/j.clinbiochem.2018.07.002. Epub 2018 Jul 6. PMID 30111510
- [Background] Karthikeyan G, Moncur RA, Levine O, Heels-Ansdell D, Chan MT, Alonso-Coello P, Yusuf S, Sessler D, Villar JC, Berwanger O, McQueen M, Mathew A, Hill S, Gibson S, Berry C, Yeh HM, Devereaux PJ. Is a pre-operative brain natriuretic peptide or N-terminal pro-B-type natriuretic peptide measurement an independent predictor of adverse cardiovascular outcomes within 30 days of noncardiac surgery? A systematic review and meta-analysis of observational studies. J Am Coll Cardiol. 2009 Oct 20;54(17):1599-606. doi: 10.1016/j.jacc.2009.06.028. PMID 19833258
- [Background] Kasahara S, Sakata Y, Nochioka K, Miura M, Abe R, Sato M, Aoyanagi H, Fujihashi T, Yamanaka S, Shiroto T, Sugimura K, Takahashi J, Miyata S, Shimokawa H. Conversion formula from B-type natriuretic peptide to N-terminal proBNP values in patients with cardiovascular diseases. Int J Cardiol. 2019 Apr 1;280:184-189. doi: 10.1016/j.ijcard.2018.12.069. Epub 2019 Jan 7. PMID 30685104
- [Background] Paniagua Iglesias P, Diaz Ruano S, Alvarez-Garcia J; VISION study collaborating researchers in Spain. Myocardial injury after noncardiac surgery. Rev Esp Cardiol (Engl Ed). 2014 Oct;67(10):794-6. doi: 10.1016/j.rec.2014.05.011. Epub 2014 Sep 7. No abstract available. PMID 25205649
- [Background] Pearse RM, Moreno RP, Bauer P, Pelosi P, Metnitz P, Spies C, Vallet B, Vincent JL, Hoeft A, Rhodes A; European Surgical Outcomes Study (EuSOS) group for the Trials groups of the European Society of Intensive Care Medicine and the European Society of Anaesthesiology. Mortality after surgery in Europe: a 7 day cohort study. Lancet. 2012 Sep 22;380(9847):1059-65. doi: 10.1016/S0140-6736(12)61148-9. PMID 22998715
- [Background] Rodseth RN, Biccard BM, Le Manach Y, Sessler DI, Lurati Buse GA, Thabane L, Schutt RC, Bolliger D, Cagini L, Cardinale D, Chong CP, Chu R, Cnotliwy M, Di Somma S, Fahrner R, Lim WK, Mahla E, Manikandan R, Puma F, Pyun WB, Radovic M, Rajagopalan S, Suttie S, Vanniyasingam T, van Gaal WJ, Waliszek M, Devereaux PJ. The prognostic value of pre-operative and post-operative B-type natriuretic peptides in patients undergoing noncardiac surgery: B-type natriuretic peptide and N-terminal fragment of pro-B-type natriuretic peptide: a systematic review and individual patient data meta-analysis. J Am Coll Cardiol. 2014 Jan 21;63(2):170-80. doi: 10.1016/j.jacc.2013.08.1630. Epub 2013 Sep 26. PMID 24076282
- [Background] Rorth R, Jhund PS, Yilmaz MB, Kristensen SL, Welsh P, Desai AS, Kober L, Prescott MF, Rouleau JL, Solomon SD, Swedberg K, Zile MR, Packer M, McMurray JJV. Comparison of BNP and NT-proBNP in Patients With Heart Failure and Reduced Ejection Fraction. Circ Heart Fail. 2020 Feb;13(2):e006541. doi: 10.1161/CIRCHEARTFAILURE.119.006541. Epub 2020 Feb 17. PMID 32065760
- [Background] Weiser TG, Regenbogen SE, Thompson KD, Haynes AB, Lipsitz SR, Berry WR, Gawande AA. An estimation of the global volume of surgery: a modelling strategy based on available data. Lancet. 2008 Jul 12;372(9633):139-144. doi: 10.1016/S0140-6736(08)60878-8. Epub 2008 Jun 24. PMID 18582931
- [Background] Nieuwkamp DJ, Algra A, Blomqvist P, Adami J, Buskens E, Koffijberg H, Rinkel GJ. Excess mortality and cardiovascular events in patients surviving subarachnoid hemorrhage: a nationwide study in Sweden. Stroke. 2011 Apr;42(4):902-7. doi: 10.1161/STROKEAHA.110.602722. Epub 2011 Feb 17. PMID 21330628
- [Result] Botto F, Alonso-Coello P, Chan MT, Villar JC, Xavier D, Srinathan S, Guyatt G, Cruz P, Graham M, Wang CY, Berwanger O, Pearse RM, Biccard BM, Abraham V, Malaga G, Hillis GS, Rodseth RN, Cook D, Polanczyk CA, Szczeklik W, Sessler DI, Sheth T, Ackland GL, Leuwer M, Garg AX, Lemanach Y, Pettit S, Heels-Ansdell D, Luratibuse G, Walsh M, Sapsford R, Schunemann HJ, Kurz A, Thomas S, Mrkobrada M, Thabane L, Gerstein H, Paniagua P, Nagele P, Raina P, Yusuf S, Devereaux PJ, Devereaux PJ, Sessler DI, Walsh M, Guyatt G, McQueen MJ, Bhandari M, Cook D, Bosch J, Buckley N, Yusuf S, Chow CK, Hillis GS, Halliwell R, Li S, Lee VW, Mooney J, Polanczyk CA, Furtado MV, Berwanger O, Suzumura E, Santucci E, Leite K, Santo JA, Jardim CA, Cavalcanti AB, Guimaraes HP, Jacka MJ, Graham M, McAlister F, McMurtry S, Townsend D, Pannu N, Bagshaw S, Bessissow A, Bhandari M, Duceppe E, Eikelboom J, Ganame J, Hankinson J, Hill S, Jolly S, Lamy A, Ling E, Magloire P, Pare G, Reddy D, Szalay D, Tittley J, Weitz J, Whitlock R, Darvish-Kazim S, Debeer J, Kavsak P, Kearon C, Mizera R, O'Donnell M, McQueen M, Pinthus J, Ribas S, Simunovic M, Tandon V, Vanhelder T, Winemaker M, Gerstein H, McDonald S, O'Bryne P, Patel A, Paul J, Punthakee Z, Raymer K, Salehian O, Spencer F, Walter S, Worster A, Adili A, Clase C, Cook D, Crowther M, Douketis J, Gangji A, Jackson P, Lim W, Lovrics P, Mazzadi S, Orovan W, Rudkowski J, Soth M, Tiboni M, Acedillo R, Garg A, Hildebrand A, Lam N, Macneil D, Mrkobrada M, Roshanov PS, Srinathan SK, Ramsey C, John PS, Thorlacius L, Siddiqui FS, Grocott HP, McKay A, Lee TW, Amadeo R, Funk D, McDonald H, Zacharias J, Villar JC, Cortes OL, Chaparro MS, Vasquez S, Castaneda A, Ferreira S, Coriat P, Monneret D, Goarin JP, Esteve CI, Royer C, Daas G, Chan MT, Choi GY, Gin T, Lit LC, Xavier D, Sigamani A, Faruqui A, Dhanpal R, Almeida S, Cherian J, Furruqh S, Abraham V, Afzal L, George P, Mala S, Schunemann H, Muti P, Vizza E, Wang CY, Ong GS, Mansor M, Tan AS, Shariffuddin II, Vasanthan V, Hashim NH, Undok AW, Ki U, Lai HY, Ahmad WA, Razack AH, Malaga G, Valderrama-Victoria V, Loza-Herrera JD, De Los Angeles Lazo M, Rotta-Rotta A, Szczeklik W, Sokolowska B, Musial J, Gorka J, Iwaszczuk P, Kozka M, Chwala M, Raczek M, Mrowiecki T, Kaczmarek B, Biccard B, Cassimjee H, Gopalan D, Kisten T, Mugabi A, Naidoo P, Naidoo R, Rodseth R, Skinner D, Torborg A, Paniagua P, Urrutia G, Maestre ML, Santalo M, Gonzalez R, Font A, Martinez C, Pelaez X, De Antonio M, Villamor JM, Garcia JA, Ferre MJ, Popova E, Alonso-Coello P, Garutti I, Cruz P, Fernandez C, Palencia M, Diaz S, Del Castillo T, Varela A, de Miguel A, Munoz M, Pineiro P, Cusati G, Del Barrio M, Membrillo MJ, Orozco D, Reyes F, Sapsford RJ, Barth J, Scott J, Hall A, Howell S, Lobley M, Woods J, Howard S, Fletcher J, Dewhirst N, Williams C, Rushton A, Welters I, Leuwer M, Pearse R, Ackland G, Khan A, Niebrzegowska E, Benton S, Wragg A, Archbold A, Smith A, McAlees E, Ramballi C, Macdonald N, Januszewska M, Stephens R, Reyes A, Paredes LG, Sultan P, Cain D, Whittle J, Del Arroyo AG, Sessler DI, Kurz A, Sun Z, Finnegan PS, Egan C, Honar H, Shahinyan A, Panjasawatwong K, Fu AY, Wang S, Reineks E, Nagele P, Blood J, Kalin M, Gibson D, Wildes T; Vascular events In noncardiac Surgery patIents cOhort evaluatioN (VISION) Writing Group, on behalf of The Vascular events In noncardiac Surgery patIents cOhort evaluatioN (VISION) Investigators; Appendix 1. The Vascular events In noncardiac Surgery patIents cOhort evaluatioN (VISION) Study Investigators Writing Group; Appendix 2. The Vascular events In noncardiac Surgery patIents cOhort evaluatioN Operations Committee; Vascular events In noncardiac Surgery patIents cOhort evaluatioN VISION Study Investigators. Myocardial injury after noncardiac surgery: a large, international, prospective cohort study establishing diagnostic criteria, characteristics, predictors, and 30-day outcomes. Anesthesiology. 2014 Mar;120(3):564-78. doi: 10.1097/ALN.0000000000000113. PMID 24534856
- [Derived] Davidson T, Parlow J, King B, DuMerton D, Roshanov PS, Devereaux PJ, Leitch J. Conversion between B-type natriuretic peptide and N-terminal pro B-type natriuretic peptide in perioperative risk assessment: protocol for a prospective cohort study. BMJ Open. 2023 May 19;13(5):e068147. doi: 10.1136/bmjopen-2022-068147. PMID 37208131